CLINICAL TRIAL: NCT01008059
Title: Novel Noninvasive Assessment of Cytochrome P4450 Activity: Simultaneous Testing Pilot
Brief Title: Alfentanil: Simultaneous Testing Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0715-201103523; 5R01GM063674-07 (NIH)
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Evaluate Two Paradigms for Simultaneous Assessment of Hepatic and Intestinal CYP3A
MeSH Terms: interventions — Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alfentanil (Experimental): Alfentanil (0.5-1 mg IV bolus) followed 3 hours later or simultaneously by 1-4 mg oral deuterium-labeled (d3) alfentanil on each study visit.
  Interventions: Drug: Alfentanil

INTERVENTIONS:
Drug: Alfentanil — No drug treatment before alfentanil

SUMMARY:
To evaluate two paradigms for simultaneous assessment of hepatic and intestinal CYP3A activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, 18-40 yr. old
* Good general health with no remarkable medical conditions such as liver, kidney, heart, or lung failure
* BMI between 20-33
* Provide informed consent

Exclusion Criteria:

* Known history of liver or kidney disease
* Use of prescription or non prescription medications, herbals or foods known to be metabolized by or affect CYP3A (including oral birth control medications)
* Females who are pregnant or nursing
* Known history of drug or alcohol addiction (prior or present addiction or treatment for addiction)
* Direct physical access to and routine handling of addicting drugs in the regular course of duty (this is a routine exclusion from studies of drugs with addiction potential).
* History of bradycardia
* Respiratory rate <10
* History of significant pulmonary disease
* History of pre-existing medical condition predisposing to respiratory depression
* Systolic blood pressure <100 mgHg and diastolic blood pressure <70mmHg

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan D Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University/Barnes Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Sequential Alfentanil: Alfentanil (IV bolus) followed 3 hours later by oral deuterium-labeled (d3) alfentanil. Control.
- Rifampin Sequential Alfentanil: Alfentanil (IV bolus) followed 3 hours later by oral deuterium-labeled (d3) alfentanil after 5d rifampin pretreatment
- Grapefruit Juice Sequential Alfentanil: Alfentanil (IV bolus) followed 3 hours later by oral deuterium-labeled (d3) alfentanil after 3 oz double strength oral grapefruit juice
- Ketoconazole Sequential Alfentanil: Alfentanil (IV bolus) followed 3 hours later by oral deuterium-labeled (d3) alfentanil after 3d ketoconazole
- Control Simultaneous Alfentanil: Alfentanil (IV bolus) and simultaneous oral deuterium-labeled (d3) alfentanil.Control.
- Rifampin Simultaneous Alfentanil: Alfentanil (IV bolus) and simultaneous oral deuterium-labeled (d3) alfentanil after 5d rifampin pretreatment
- Grapefruit Juice Simultaneous Alfentanil: Alfentanil (IV bolus) and simultaneous oral deuterium-labeled (d3) alfentanil after 3 oz double strength oral grapefruit juice
- Ketoconazole Simultaneous Alfentanil: Alfentanil (IV bolus) and simultaneous oral deuterium-labeled (d3) alfentanil after 3d ketoconazole
Period: Control Sequential Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Rifampin Sequential Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Grapefruit Juice Sequential Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Ketoconazole Sequential Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Control Simultaneous Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Rifampin Simultaneous Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Grapefruit Juice Simultaneous Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Ketoconazole Simultaneous Alfentanil
Arm/Group | Control Sequential Alfentanil | Rifampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alfentanil
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Alfentanil Concentration vs. Time Extrapolated to Infinity
Description: AUC(0-inf)
Time Frame: 9 hours
Measure: Mean (Standard Deviation); unit: (hr*ng/ml/mg)
Arm/Group | Alfentanil
Number analyzed (Participants) | 6
(hr*ng/ml/mg)
  Simultaneous Control | 58 (15)
  Simultaneous Rifampin | 57 (9)
  Simultaneous Grapefruit | 55 (12)
  Simultaneous ketoconazole | 73 (26)
  Sequential Control | 59 (27)
  Sequential Rifampin | 54 (10)
  Sequential Grapefruit | 59 (31)
  Sequential Ketoconazole | 73 (19)
Statistical Analysis 1: Comparison: Alfentanil; Test type: Superiority; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Refampin Sequential Alfentanil: Alfentanil (IV bolus) followed 3 hours later by oral deuterium-labeled (d3) alfentanil after 5d rifampin pretreatment
Arm/Group | Control Sequential Alfentanil | Refampin Sequential Alfentanil | Grapefruit Juice Sequential Alfentanil | Ketoconazole Sequential Alfentanil | Control Simultaneous Alfentanil | Rifampin Simultaneous Alfentanil | Grapefruit Juice Simultaneous Alfentanil | Ketoconazole Simultaneous Alfentanil
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Sequential Alfentanil (N=6) | Refampin Sequential Alfentanil (N=6) | Grapefruit Juice Sequential Alfentanil (N=6) | Ketoconazole Sequential Alfentanil (N=6) | Control Simultaneous Alfentanil (N=6) | Rifampin Simultaneous Alfentanil (N=6) | Grapefruit Juice Simultaneous Alfentanil (N=6) | Ketoconazole Simultaneous Alfentanil (N=6)
Nausea/Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes